CLINICAL TRIAL: NCT02782585
Title: Hypoalgesic Effects of Three Different Manual Therapy Techniques on Cervical Spine and Psychological Interaction: Randomized Clinical Trial
Brief Title: Manual Therapy Techniques on Cervical Spine and Psychological Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Psychological interaction
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Neck Pain
Keywords: neck pain; Manual therapy; psychological interaction
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental group 1 (Experimental): Cervical Manipulation
  Interventions: Other: Cervical manipulation
- Experimental group 2 (Experimental): Cervical lateral glide
  Interventions: Other: Cervical lateral glide
- Control group (Placebo Comparator): Cervical Mobilisation
  Interventions: Other: Cervical mobilisation

INTERVENTIONS:
Other: Cervical manipulation — The therapist cradled the subject´s head with the other hand. Gentle ipsilateral side flexion and contralateral rotation to the targeted side were introduced until slight tension was perceived in the tissues at the contact point. The High velocity, low amplitude (HVLA) manipulation was directed upward and medially in the direction of the subject´s contralateral eye. The therapist monitored for cavitation or 'popping sound' accompanying the manipulations. If an audible popping sound was not heard during the first manipulative attempt, the procedure was repeated in the second time.
  Arms: Experimental group 1
Other: Cervical lateral glide — The upper limb of the right side of subjects was maintained in rest, with the arm along the trunk and the hand over the abdominal wall. The right hand of the treating therapist was positioned over scapula region, to depress the scapula while left hand cradled the occiput and neck above C5-C6 and left hand produced a passive lateral movement of the occipital and neck region.
  Arms: Experimental group 2
Other: Cervical mobilisation — The patients received a passive cervical mobilization that involved a grade III oscillatory unilateral posteroanterior mobilization to the right articular pillar of C5/C6 segment as described Maitland at a frequency of 2Hz. All the subjects were positioned in prone position as the protocol described by Sterling et al. for 3 sets of 2 minutes with 1 minute rest between sets.
  Arms: Control group

SUMMARY:
Manual therapy (MT) techniques applied over cervical region have over both local (neck) and distant regions (elbow) in both asymptomatic and symptomatic populations. Neurophysiological mechanisms are hypothesized to explain the underlying effects, with effects originating from peripheral mechanisms, spinal cord and supraspinal mechanisms.

There is also an increasing interest in the study of the role of psychological variables in the treatment success in neck pain. Psychological variables, like anxiety catastrophizing or kinesiophobia are related to poor prognosis in the development of pain outcomes and disability in neck pain, being the Fear-Avoidance Model of pain one of the most tested models in this field.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain

Exclusion Criteria:

* myelopathy
* fracture
* infection
* dystonia
* tumor
* inflammatory disease
* fibromyalgia
* or osteoporosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from Pressure Pain Thresholds (PPT) at 24 hours | 24 hours, 5 minutes after the treatment
  PPT will be assessed bilaterally over the C7 zygapophyseal joint, epicondyle region, and trapezious muscle by an assessor blinded to the subjects condition.
Change from State-Trait Anxiety Inventory subscale (STAI-E) at 24 hours | 24 hours, 5 minutes after the treatment
  Will be used to measure anxiety status

SECONDARY OUTCOMES:
Beck depression Inventory (BDI-II) | 24 hours, 5 minutes after the treatment
  Will be used to measure depression status
Tampa Scale for Kinesiophobia | 24 hours, 5 minutes after the treatment
  Will be used to measure Kinesiophobia status

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alonso-Perez JL, Lopez-Lopez A, La Touche R, Lerma-Lara S, Suarez E, Rojas J, Bishop MD, Villafane JH, Fernandez-Carnero J. Hypoalgesic effects of three different manual therapy techniques on cervical spine and psychological interaction: A randomized clinical trial. J Bodyw Mov Ther. 2017 Oct;21(4):798-803. doi: 10.1016/j.jbmt.2016.12.005. Epub 2016 Dec 22. PMID 29037630